CLINICAL TRIAL: NCT07240493
Title: Evaluating the Effect of Bone Morphogenetic Protein on Dental Implant Stability and Marginal Bone Level Following Immediate Implant Placement (Randomized Controlled Study)
Brief Title: BMP Effect on Implant Stability and Marginal Bone Level After Immediate Placement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Adil Saeed (Other)
Responsible Party: Sponsor-Investigator, Aya Adil Saeed, principal investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 991124
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Unrestorable Tooth Replaced by Immediate Implant With BMP

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: rhBMP-2 Group (Experimental): Immediate dental implant placement with application of recombinant human Bone Morphogenetic Protein-2 (rhBMP-2) with bone graft in jumping gap.
  Interventions: Biological: rhBMP-2 placement
- Control: standard immediate implant (Active Comparator): Standard immediate dental implant placement procedure without application of Bone Morphogenetic Protein.
  Interventions: Device: conventional immediate implant

INTERVENTIONS:
Biological: rhBMP-2 placement — rhBMP-2 is mixed with BCP bone graft and placed in the jumping gap after immediate dental implant placement.
  Arms: Experimental: rhBMP-2 Group
Device: conventional immediate implant — Standard immediate dental implant placement procedure without adding of Bone Morphogenetic Protein in the bone graft placed in the jumping gap.
  Arms: Control: standard immediate implant

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effect of recombinant human Bone Morphogenetic Protein-2 (rhBMP-2) on the stability and marginal bone level of dental implants following immediate placement.

patients requiring extraction of unrestorable tooth in upper incisors or premolar region will be randomly assigned into two groups: the experimental group will receive immediate implant placement with rhBMP-2 application, while the control group will receive immediate implant placement without rhBMP-2.

each group includes 16 immediate implants. Implant stability will be assessed using resonance frequency analysis (RFA) at baseline, and 16 weeks after implant placement. Marginal bone level changes will be evaluated radiographically using cone beam computed tomography (CBCT).

The study aims to determine whether the use of rhBMP-2 enhances osseointegration and reduces marginal bone loss compared with conventional immediate implant placement.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy patients ≥18 years of either sex, having a single or multiple unrestorable maxillary anterior and premolar teeth which are indicated for extraction, where a jumping gap is most likely to form (≥2mm) provides a reliable environment to study the local effects of rhBMP-2 in consistent and replicable conditions.

  2. Apical bone ≥ 3mm from the vertical structure showed in x-rays beyond the apex.

  3. Patients who are willing to comply the study and agree to provide their consent.

  4. Good to fair oral hygiene.

Exclusion Criteria:

- 1. Active infection or inflammation in implant area. 2. Medically compromised patients such as uncontrolled diabetes, coagulation disorders, immune compromised patient, patient treated with bisphosphate drugs, psychiatric problems, pregnant women, or any medical condition that affect bone healing.

3. Clinical evidence of parafunctional habits. 4. Heavy smokers (≥20 cigarettes a day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Implant Stability Quotient (ISQ) measured by Resonance Frequency Analysis | Baseline and 16 weeks after implant placement
  Evaluation of implant stability using resonance frequency analysis (RFA) device to measure the Implant Stability Quotient (ISQ) at baseline and 16 weeks after implant placement.

SECONDARY OUTCOMES:
Marginal Bone Level (MBL) Changes around Dental Implants | Baseline and 16 weeks after implant placement
  Radiographic assessment of marginal bone level (MBL) around dental implants using Cone Beam Computed Tomography (CBCT) at baseline and 16 weeks after implant placement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad - College of Dentistry, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is an academic clinical study with a limited number of participants, and data will be used only for internal analysis within the University of Baghdad.